CLINICAL TRIAL: NCT02281435
Title: One-arm, Open Label, Phase I (Out of 3 Phases), Pilot Study to Verify the Safety of PrePex™ Device for Screen Failure Subjects (Men With Narrow Foreskin and Phimosis) for Adult Male Circumcision, Performed by Physicians, in a Male Population That is Scheduled to Undergo Circumcision in an Effort to Prevent the Spread of HIV.
Brief Title: Follow Up Study to Evaluate a Non-Surgical Device for Adult Male Circumcision for Screen Failure Subjects
Acronym: RMC-05
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Rwanda (Other Government)
Responsible Party: Principal Investigator, Vincent Mutabazi, Director of the Research Grants Unit, Ministry of Health, Rwanda
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RMC-05 (Phase I)
Record Dates: First submitted 2014-05-22; First posted 2014-11-03 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Male Circumcision; HIV Prevention; Screen Failure Subjects; Narrow Foreskin
Keywords: Male Circumcision; HIV Prevention; Screen Failure Subjects; PrePex with Incision

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PrePex with Incision (Experimental): Adult male circumcision by the PrePex™ device using foreskin incision
  Interventions: Device: PrePex™ device

INTERVENTIONS:
Device: PrePex™ device — PrePex™ device for adult male circumcision. The PrePex™ device facilitates adult male circumcision that is bloodless with no anesthesia and no sutures, but in this study the procedure consist an incision on to the foreskin.

SUMMARY:
It is well known from a range of observational and epidemiological studies that the lifetime risk of acquiring HIV among males can be significantly reduced via circumcision by 53%-60% and by up to 73% in post-trial observation. Numerous papers on the topic have been published over the past two decades to elevate HIV prevention awareness, especially in sub-Saharan countries.

Results from the Decision Makers' Program Planning Tool (DMPPT) models, performed in 2011, suggest that scaling up adult voluntary medical male circumcision (VMMC) to reach 80% coverage in the 13 countries by 2015 would entail performing 20.34 million circumcisions between 2011 and 2015 and additional 8.42 million between 2016 and 2025. Such a scale-up would result in averting 3.36 million new HIV infections through 2025. In addition, while the model shows that this scale-up would cost a total of US$2 billion between 2011 and 2025, it would result in net savings (due to averted treatment and care costs) amounting to US$16.51 billion.

To date, there are over 38 million adolescent and adult males in Africa that could benefit from male circumcision (MC) for HIV prevention. The challenge Africa faces is how to safely scale up a surgical procedure in resource limited settings.

DETAILED DESCRIPTION:
Rwanda has a national plan to offer a Voluntary Medical Male Circumcision (VMMC) program to 2 million adult men in 2 years as part of a comprehensive HIV prevention strategy.

The PrePex device was granted with pre-qualification approval on May 2013 by the World Health Organization (WHO), for scaling up VMMC in Africa.

The device works by stopping the flow of blood to the distal foreskin, leading to necrosis of the tissue, which is removed with the device after 7 days.

The PrePex device was developed to facilitate rapid scale up of non-surgical adult male circumcision in resource limited settings, and it is the first MC device which was granted with a WHO recommendation in addition to CE and FDA approvals.

Prior studies showed that between 8%-12% of men are contraindicated for the standard PrePex technique due to very narrow foreskin from border cases to severe Phimosis, preventing insertion of the Inner Ring of the PrePex device.

The main objective of the study was to test the safety of a new male circumcision technique, using the same PrePex device (PrePex with incision). The new technique entails the use of local anesthesia and thereafter an incision in the foreskin. PrePex with incision technique was planned to allow PrePex non-surgical contraindicated patients to undergo VMMC with the device, thus avoiding conventional surgery and suturing. The study also included analysis of potential benefits the PrePex with incision technique has over conventional surgical circumcision.

The study has 3 phases, the current results represent Phase I - testing the feasibility and safety of the PrePex with incision procedure, intended to screen failure subjects of the standard PrePex procedure. Phase I includes performing feasibility testing on 6 subjects using 2 different techniques and once feasibility is demonstrated to include an additional Analysis phase of data collection from additional 30 subjects to reinforce the safety of the one chosen technique.

Phase II will includes a special non-surgical PrePex procedure for patients with narrow foreskin that will entail the usage of Lidocaine anesthetic cream 30 minutes pre procedure and additional force in inserting of the Inner Ring (hereto: Special PrePex procedure).

Phase III will includes performing additional PrePex with incision procedures with local anesthesia and special PrePex procedure incision to achieve a statistical significant sample size and determine the recommended guideline and procedure for performing PrePex on men with narrow foreskin and phimosis.

ELIGIBILITY:
Inclusion Criteria:

* Ages - 21 to 49 years
* Subject wants to be circumcised
* Uncircumcised
* HIV sero-negative
* Able to understand the study procedures and requirements
* Agrees to abstain sexual intercourse for 9 weeks
* Agrees to abstain from masturbation for 2 weeks
* Agrees to remain in the health care facility for up to 48 hours post procedure as required
* Agrees to return to the health care facility for follow-up visits (or as instructed) after his circumcision for a period of 8 weeks post removal (9 weeks total)
* Subject able to comprehend and freely give informed consent for participation in this study and is considered by the investigator to have good compliance for the study
* Subject agrees to anonymous video and photographs of the procedure and follow up visits
* Subject that was a medical screen failure in RMC-03 study.

Exclusion Criteria:

* Active genital infection, anatomic abnormality or other condition, which in the opinion of the investigator prevents the subject from undergoing circumcision according to the study procedure and can only undergo surgical MC
* HIV sero-positive
* Known bleeding / coagulation abnormality, uncontrolled diabetes
* Subject does not agree to anonymous video and photographs of the procedure and follow up visits
* Refusal to take HIV test
* Refuse to be hospitalized in the medical center for up to 48 hours post Placement as required
* Subjects that should be excluded from standard surgical MC, such as warts under the prepuce, hypospadias, epispadias, un treated UTI.

Ages: 21 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Rate of clinical Adverse Events (AEs) | 11 months
  To verify that the incidence of moderate and severe Clinical AEs and device-related Adverse Events are not significantly higher than 2%.

SECONDARY OUTCOMES:
Rate of complete circumcision | 11 months
  Glans fully exposed
Time to complete healing | 11 months
  Average time to complete healing
Device related incidents | 11 months
  Necrotic Process not initiated, i.e the device does not perform according to its intended use of stopping blood flow to the foreskin.
  o Device does not remain in situ. (a case where subject is not compliance with counseling instructions and actively moves the device from its place, will not be considered a device related incident)
Optimal methodology to perform PrePex procedure on subjects with very narrow opening of the foreskin. | 11 months
  Technique 1 Vs. technique 2
Safety and effectiveness of performing PrePex MC for subjects with tight frenulum or torn frenulum | 11 months
  Device safety was assessed by the rate of clinical adverse events and device-related incidents.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Mutabazi, M.D., Principal Investigator — Ministry of Health, Rwanda; Jean Paul Bitega, M.D., Principal Investigator — Rwanda Military Hospital
Locations (1):
- Rwanda Military Hospital, Kigali, Rwanda

REFERENCES:
- See also: Rwanda Biomedical Centre — http://www.rbc.gov.rw/